CLINICAL TRIAL: NCT02575235
Title: Randomized, Double Blinded, Placebo-controlled Trial to Assess the Preventive Effects of Cetylpyridinium Chloride on Sarcopenia
Brief Title: Clinical Trial to Assess the Preventive Effects of Cetylpyridinium Chloride on Sarcopenia
Acronym: CPC2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNUHRM-CPC2
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Cetylpyridinium chloride
MeSH Terms: conditions — Sarcopenia | interventions — Cetylpyridinium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.5mg Cetylpyridinium Chloride (CPC) (Experimental): 1.5mg CPC will be taken daily for four weeks.
  Interventions: Drug: Cetylpyridinium Chloride (CPC)
- 4.5mg Cetylpyridinium Chloride (CPC) (Experimental): 4.5mg CPC will be taken daily for four weeks.
  Interventions: Drug: Cetylpyridinium Chloride (CPC)
- Control (Placebo Comparator): Placebo will be taken daily for four weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cetylpyridinium Chloride (CPC) — Two study groups take CPC of 1.5mg and 4.5mg daily for four weeks.
  Arms: 1.5mg Cetylpyridinium Chloride (CPC); 4.5mg Cetylpyridinium Chloride (CPC)
Drug: placebo — Control group takes the placebo for the same period.
  Arms: Control

SUMMARY:
This study is to assess the impact on the prevention of sarcopenia after taking cetylpyridinium chloride targeting the patients of pre-sarcopenia or sarcopenia over the age of 60

DETAILED DESCRIPTION:
75 people that meet the inclusion criteria on screening test are assigned to one of three groups by randomization. They take the medication for four weeks under doubleblind. Two study groups take cetylpyridinium chloride of 1.5mg, 4.5mg daily for four weeks. Control group takes the placebo for the same period. The main outcome variables are measured and compared respectively in baseline, immediately after dosing end and two weeks, four weeks after the end of administration. Finally cetylpyridinium chloride is verified whether it has a preventive effect on sarcopenia and set an appropriate dose.

ELIGIBILITY:
Inclusion Criteria:

* Pre-sarcopenia A. Reduced skeletal muscle mass (appendicular skeletal muscle mass/height2) M < 7.0kg/m2, F < 5.7kg/m2

Exclusion Criteria:

* History of stroke or spinal cord injury
* Artificial joint
* Acute disease or unstable chronic disease
* Phenylketonuria
* History of myocardiac infarction
* Allergic contact dermatitis
* History of drug/alcohol addiction, habitual smoker

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in procollagen type III N-terminal peptide | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration

SECONDARY OUTCOMES:
Change from baseline in insulin like growth factor 1 (IGF-1) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in transforming growth factor β1 (TGF-β1) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in Myostatin | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in tumor necrosis factor α (TNF-α) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in interleukin 1 (IL-1) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in fatty acid binding protein 3 (FABP3) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in monocyte chemoattractant protein 1 (MCP-1) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in Skeletal muscle index | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in short physical performance battery (SPPB) | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration
Change from baseline in Grip strength | baseline, two weeks after administration start, immediately after dosing end, two weeks after the end of administration, four weeks after the end of administration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Pahor M, Manini T, Cesari M. Sarcopenia: clinical evaluation, biological markers and other evaluation tools. J Nutr Health Aging. 2009 Oct;13(8):724-8. doi: 10.1007/s12603-009-0204-9. PMID 19657557
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Hong S, Oh HJ, Choi H, Kim JG, Lim SK, Kim EK, Pyo EY, Oh K, Kim YT, Wilson K, Choi WH. Characteristics of body fat, body fat percentage and other body composition for Koreans from KNHANES IV. J Korean Med Sci. 2011 Dec;26(12):1599-605. doi: 10.3346/jkms.2011.26.12.1599. Epub 2011 Nov 29. PMID 22147997
- [Background] Kalyani RR, Corriere M, Ferrucci L. Age-related and disease-related muscle loss: the effect of diabetes, obesity, and other diseases. Lancet Diabetes Endocrinol. 2014 Oct;2(10):819-29. doi: 10.1016/S2213-8587(14)70034-8. Epub 2014 Mar 6. PMID 24731660
- [Background] Ormsbee MJ, Prado CM, Ilich JZ, Purcell S, Siervo M, Folsom A, Panton L. Osteosarcopenic obesity: the role of bone, muscle, and fat on health. J Cachexia Sarcopenia Muscle. 2014 Sep;5(3):183-92. doi: 10.1007/s13539-014-0146-x. Epub 2014 Apr 17. PMID 24740742
- [Background] Moller N, Vendelbo MH, Kampmann U, Christensen B, Madsen M, Norrelund H, Jorgensen JO. Growth hormone and protein metabolism. Clin Nutr. 2009 Dec;28(6):597-603. doi: 10.1016/j.clnu.2009.08.015. Epub 2009 Sep 20. PMID 19773097
- [Background] Miller MD, Crotty M, Giles LC, Bannerman E, Whitehead C, Cobiac L, Daniels LA, Andrews G. Corrected arm muscle area: an independent predictor of long-term mortality in community-dwelling older adults? J Am Geriatr Soc. 2002 Jul;50(7):1272-7. doi: 10.1046/j.1532-5415.2002.50316.x. PMID 12133024
- [Background] Enoki H, Kuzuya M, Masuda Y, Hirakawa Y, Iwata M, Hasegawa J, Izawa S, Iguchi A. Anthropometric measurements of mid-upper arm as a mortality predictor for community-dwelling Japanese elderly: the Nagoya Longitudinal Study of Frail Elderly (NLS-FE). Clin Nutr. 2007 Oct;26(5):597-604. doi: 10.1016/j.clnu.2007.06.008. Epub 2007 Jul 31. PMID 17669559
- [Background] Stephen WC, Janssen I. Sarcopenic-obesity and cardiovascular disease risk in the elderly. J Nutr Health Aging. 2009 May;13(5):460-6. doi: 10.1007/s12603-009-0084-z. PMID 19390754
- [Background] Rolland Y, Czerwinski S, Abellan Van Kan G, Morley JE, Cesari M, Onder G, Woo J, Baumgartner R, Pillard F, Boirie Y, Chumlea WM, Vellas B. Sarcopenia: its assessment, etiology, pathogenesis, consequences and future perspectives. J Nutr Health Aging. 2008 Aug-Sep;12(7):433-50. doi: 10.1007/BF02982704. PMID 18615225
- [Background] Landi F, Marzetti E, Martone AM, Bernabei R, Onder G. Exercise as a remedy for sarcopenia. Curr Opin Clin Nutr Metab Care. 2014 Jan;17(1):25-31. doi: 10.1097/MCO.0000000000000018. PMID 24310054
- [Background] Adamo ML, Farrar RP. Resistance training, and IGF involvement in the maintenance of muscle mass during the aging process. Ageing Res Rev. 2006 Aug;5(3):310-31. doi: 10.1016/j.arr.2006.05.001. Epub 2006 Sep 1. PMID 16949353
- [Background] Morley JE, Malmstrom TK. Frailty, sarcopenia, and hormones. Endocrinol Metab Clin North Am. 2013 Jun;42(2):391-405. doi: 10.1016/j.ecl.2013.02.006. PMID 23702408
- [Background] Dalton JT, Barnette KG, Bohl CE, Hancock ML, Rodriguez D, Dodson ST, Morton RA, Steiner MS. The selective androgen receptor modulator GTx-024 (enobosarm) improves lean body mass and physical function in healthy elderly men and postmenopausal women: results of a double-blind, placebo-controlled phase II trial. J Cachexia Sarcopenia Muscle. 2011 Sep;2(3):153-161. doi: 10.1007/s13539-011-0034-6. Epub 2011 Aug 2. PMID 22031847
- [Background] White HK, Petrie CD, Landschulz W, MacLean D, Taylor A, Lyles K, Wei JY, Hoffman AR, Salvatori R, Ettinger MP, Morey MC, Blackman MR, Merriam GR; Capromorelin Study Group. Effects of an oral growth hormone secretagogue in older adults. J Clin Endocrinol Metab. 2009 Apr;94(4):1198-206. doi: 10.1210/jc.2008-0632. Epub 2009 Jan 27. PMID 19174493
- [Background] Kuang S, Rudnicki MA. The emerging biology of satellite cells and their therapeutic potential. Trends Mol Med. 2008 Feb;14(2):82-91. doi: 10.1016/j.molmed.2007.12.004. Epub 2008 Jan 22. PMID 18218339
- [Background] Kunkel SD, Elmore CJ, Bongers KS, Ebert SM, Fox DK, Dyle MC, Bullard SA, Adams CM. Ursolic acid increases skeletal muscle and brown fat and decreases diet-induced obesity, glucose intolerance and fatty liver disease. PLoS One. 2012;7(6):e39332. doi: 10.1371/journal.pone.0039332. Epub 2012 Jun 20. PMID 22745735
- [Background] Narkar VA, Downes M, Yu RT, Embler E, Wang YX, Banayo E, Mihaylova MM, Nelson MC, Zou Y, Juguilon H, Kang H, Shaw RJ, Evans RM. AMPK and PPARdelta agonists are exercise mimetics. Cell. 2008 Aug 8;134(3):405-15. doi: 10.1016/j.cell.2008.06.051. Epub 2008 Jul 31. PMID 18674809
- [Background] Harrison DE, Strong R, Sharp ZD, Nelson JF, Astle CM, Flurkey K, Nadon NL, Wilkinson JE, Frenkel K, Carter CS, Pahor M, Javors MA, Fernandez E, Miller RA. Rapamycin fed late in life extends lifespan in genetically heterogeneous mice. Nature. 2009 Jul 16;460(7253):392-5. doi: 10.1038/nature08221. Epub 2009 Jul 8. PMID 19587680
- [Background] Potsch MS, Tschirner A, Palus S, von Haehling S, Doehner W, Beadle J, Coats AJ, Anker SD, Springer J. The anabolic catabolic transforming agent (ACTA) espindolol increases muscle mass and decreases fat mass in old rats. J Cachexia Sarcopenia Muscle. 2014 Jun;5(2):149-58. doi: 10.1007/s13539-013-0125-7. Epub 2013 Nov 22. PMID 24272787
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Chien MY, Huang TY, Wu YT. Prevalence of sarcopenia estimated using a bioelectrical impedance analysis prediction equation in community-dwelling elderly people in Taiwan. J Am Geriatr Soc. 2008 Sep;56(9):1710-5. doi: 10.1111/j.1532-5415.2008.01854.x. Epub 2008 Aug 6. PMID 18691288
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Lauretani F, Russo CR, Bandinelli S, Bartali B, Cavazzini C, Di Iorio A, Corsi AM, Rantanen T, Guralnik JM, Ferrucci L. Age-associated changes in skeletal muscles and their effect on mobility: an operational diagnosis of sarcopenia. J Appl Physiol (1985). 2003 Nov;95(5):1851-60. doi: 10.1152/japplphysiol.00246.2003. PMID 14555665
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Reagan-Shaw S, Nihal M, Ahmad N. Dose translation from animal to human studies revisited. FASEB J. 2008 Mar;22(3):659-61. doi: 10.1096/fj.07-9574LSF. Epub 2007 Oct 17. PMID 17942826
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Bhasin S, He EJ, Kawakubo M, Schroeder ET, Yarasheski K, Opiteck GJ, Reicin A, Chen F, Lam R, Tsou JA, Castaneda-Sceppa C, Binder EF, Azen SP, Sattler FR. N-terminal propeptide of type III procollagen as a biomarker of anabolic response to recombinant human GH and testosterone. J Clin Endocrinol Metab. 2009 Nov;94(11):4224-33. doi: 10.1210/jc.2009-1434. Epub 2009 Oct 16. PMID 19837911
- [Background] Chen F, Lam R, Shaywitz D, Hendrickson RC, Opiteck GJ, Wishengrad D, Liaw A, Song Q, Stewart AJ, Cummings CE, Beals C, Yarasheski KE, Reicin A, Ruddy M, Hu X, Yates NA, Menetski J, Herman GA. Evaluation of early biomarkers of muscle anabolic response to testosterone. J Cachexia Sarcopenia Muscle. 2011 Mar;2(1):45-56. doi: 10.1007/s13539-011-0021-y. Epub 2011 Feb 26. PMID 21475673
- [Background] Moerman DE, Jonas WB. Deconstructing the placebo effect and finding the meaning response. Ann Intern Med. 2002 Mar 19;136(6):471-6. doi: 10.7326/0003-4819-136-6-200203190-00011. PMID 11900500
- [Background] Lopez-Gomez M, Corona T, Diaz-Ruiz A, Rios C. Safety and tolerability of dapsone for the treatment of patients with drug-resistant, partial-onset seizures: an open-label trial. Neurol Sci. 2011 Dec;32(6):1063-7. doi: 10.1007/s10072-011-0612-6. Epub 2011 May 17. PMID 21584739
- [Background] Damodar S, Viswabandya A, George B, Mathews V, Chandy M, Srivastava A. Dapsone for chronic idiopathic thrombocytopenic purpura in children and adults--a report on 90 patients. Eur J Haematol. 2005 Oct;75(4):328-31. doi: 10.1111/j.1600-0609.2005.00545.x. PMID 16146539
- [Background] Sharquie KE, Najim RA, Abu-Raghif AR. Dapsone in Behcet's disease: a double-blind, placebo-controlled, cross-over study. J Dermatol. 2002 May;29(5):267-79. doi: 10.1111/j.1346-8138.2002.tb00263.x. PMID 12081158